

| BI Study Number: | 1237-0109 |
|---|---|
| Title: | Safety profile of Tiotropium + Olodaterol used as maintenance treatment in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data |
| NCT number: | NCT05393245 |
| Date: | 03 Nov 2022 |

This page has been added to the Statistical and Epidemiological Analysis Plan (SEAP) to reflect the requirements by ClinicalTrials.gov. This information is not part of the standard document.



# STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP) FOR NON-INTERVENTIONAL STUDIES (NIS)

| Γ | |
|---|---|
| Document Number: | c40431892 -01 |
| BI Study Number: | 1237-0109 |
| BI Investigational<br>Product(s) | Spiolto Respimat |
| Title: | Safety profile of Tiotropium + Olodaterol used as maintenance treatment in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data |
| Brief lay title: | Safety of Tiotropium + Olodaterol in COPD patients in Taiwan:<br>a non-interventional study based on the Taiwan National Health<br>Insurance (NHI) data |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | Not applicable |
| NIS Statistician [SEAP author] | The SEAP is prepared by the principal investigator, an epidemiologist, but not a statistician. |
| NIS Lead [SEAP reviewer] | |
| NIS Data Manager<br>[SEAP reviewer] | |
| @ 2022 | Proprietary confidential information |

© 2022 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

001-MCS-90-118\_RD-20 (2.0) / Saved on: 03 Feb 2021

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **TABLE OF CONTENTS**

| TITLE | E PAGE | . 1 |
|-------|--------------------------------------------------|-----|
| TABL | E OF CONTENTS | 2 |
| 1. I | LIST OF ABBREVIATIONS | 3 |
| 2. I | RESPONSIBLE PARTIES | 3 |
| 3. I | PURPOSE AND SCOPE | 4 |
| 4. | AMENDMENTS AND UPDATES | 5 |
| 5. I | RESEARCH QUESTION AND OBJECTIVE | 5 |
| 6. I | RESEARCH METHODS | 5 |
| 6.1 | STUDY DESIGN | - |
| 6.2 | SETTING | |
| 6.3 | STUDY POPULATION | |
| 6.4 | STUDY VISITS | |
| | VARIABLES | |
| 7.1 | EXPOSURES | |
| 7.2 | OUTCOMES | |
| | 2.1 Primary outcomes | |
| /.2 | 2.2 Secondary outcomes | 11 |
| 7.3 | COVARIATES | 1 2 |
| | DATA SOURCES | |
| | DATA MANAGEMENT AND SOFTWARE/TOOLS | |
| 9.1 | SOFTWARE/TOOLS | |
| 9.1 | HANDLING OF MISSING VALUES | |
| 9.3 | HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS | |
| | DATA ANALYSIS | |
| 10.1 | MAIN ANALYSIS | |
| 10.3 | SAFETY ANALYSIS | 17 |
| 11. ( | QUALITY CONTROL | 17 |
| | REFERENCES | |
| | PUBLISHED REFERENCES. | |
| 12.2 | UNPUBLISHED REFERENCES | 18 |
| ANNE | EX 1. ADDITIONAL INFORMATION | 19 |
| ANNE | EX 2. REVIEWERS AND APPROVAL SIGNATURES | 38 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. LIST OF ABBREVIATIONS

AE Adverse Event

BI Boehringer Ingelheim CI Confidence Interval

COPD Chronic Obstructive Pulmonary Disease

DMRP Data management and review plan

FDC Fixed dose combination ICS Inhaled corticolsteroids IQR Interquartile range

LABA Long-acting β2-agonists

LAMA Long-acting muscarinic antagonists
NHI Taiwan National Health Insurance

NHIRD Taiwan National Health Insurance Research Database

NIS Non-interventional study

Olo Olodaterol

SAE Serious Adverse Event

SEAP Statistical and epidemiological analysis plan

Tio Tiotropium

#### 2. RESPONSIBLE PARTIES

NIS Statistician [SEAP author]: , the principal investigator who is an epidemiologist and not a statistician

#### SEAP reviewers are:

- BI NIS Lead [SEAP reviewer] (in all cases):
- NIS Data Manager [SEAP reviewer] (in all cases): @!20210208
- RWE CoE [SEAP reviewer] (for all globally initiated studies and for local studies) involving BI products and Global NIS not involving BI products:
- TSTAT (for NISnd only): NA
- TM Epi [SEAP reviewer] (When BI NIS lead is not TM Epi; in all cases):

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. PURPOSE AND SCOPE

According to requirement by local regulatory authority, the safety information of newly approved drugs is to be collected to provide supplementary data to those identified in randomized clinical studies within 5 years period after approval. This is a non-interventional study based on existing data. It will provide the safety information of Spiolto (tiotropium+olodaterol) in Chinese patients with chronic obstructive pulmonary disease (COPD) in routine clinical practice in Taiwan.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. AMENDMENTS AND UPDATES

None

### 5. RESEARCH QUESTION AND OBJECTIVE

#### Primary objective:

• To estimate the incidence rate of safety outcomes in patients with COPD who initiated Tio/Olo between 1st January 2014 and 31st December 2019;

#### Secondary objective:

• To compare the baseline characteristics of patients between those treated with Tio/Olo and those with other LAMA/LABAs FDC (Vilanterol/Umeclidinium; Indacaterol /Glycopyrronium) or (LABA: Salmeterol; Formoterol; Procaterol; Indacaterol; Olodaterol, LAMA: Tiotropium bromide; Glycopyrrolate; Umeclidinium) free combination;

#### 6. RESEARCH METHODS

#### 6.1 STUDY DESIGN

This study will be a non-interventional cohort study using Taiwan National Health Insurance (NHI) claims database, Taiwan Cancer Registry (TCR) and Taiwan Mortality Data. It is a secondary health data environment with relevant information on treatment and disease outcomes of COPD patients among a population of predominantly ethnic Han Chinese. As a publicly funded single payor health insurance program, a wide range health services, including hospital care, emergency visits, ambulatory clinic services, and prescription drugs are covered for virtually all Taiwan residents. The complete capture of health care encounters reimbursed by NHI among a defined group of patients has served as the basis of many longitudinal studies that evaluated safety profiles of prescribed medications.

Health data that are available for research are provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, Ministry of Health and Welfare. The HWDSC staff encrypt the national ID for all individuals according to a secure encryption algorithm that is specific for each study, and the encrypted ID all individuals is used for linkage between databases. While the study will provide safety data on drugs of interest, from a regulatory perspective the source data are not auditable, nor de-identified individual level data be brought outside of HWDSC for independent verification of analysis.

Limitations of health insurance databases are well-known, as there is no information on results of clinical parameters (such as blood pressure and body mass index), clinical examinations (such as spirometry findings), or life style attributes (such as smoking). A

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

specific items that needs to be considered for this particular study project is whether the findings are generalizable to COPD patients in China. While there is high similarity between COPD patients in Taiwan and those in China in terms of ethnicity and dietary patterns, management patterns for COPD patients, including comorbid conditions, concomitant medications, and use of traditional Chinese medication regimens, may be different.

Taking into account the strengths and potential limitations of the data source, the population-based nature and potentially large study size of patients on drugs of interest are the major reasons that this data source is a viable option for the study.

#### 6.2 SETTING

Data used in this study will come from the Taiwan National Health Insurance (NHI) claims data. Cohort for incident Tio/Olo combined inhaler use would be identified from 2014 through 2019, with a 1-year look-back period to define new user. Cohort for other incident LAMA/LABAs combined inhaler use would be identified from 2014 through 2019, and also with a 1-year look-back period to define new user.

#### 6.3 STUDY POPULATION

#### For incident Tio/Olo combined inhaler cohort

#### • Inclusion criteria:

- 1. At least one prescription for Tio+Olo (fixed dose combination (FDC) or free combination) as a new initiation between 1<sup>st</sup> January 2014 and 31<sup>st</sup> December 2019 (the free combination will be defined as the prescriptions of the two compounds on the same day);
- 2. Aged ≥ 40 years on the index date (The first dispensing of Tio+Olo combined inhaler will be defined as the index date);
- 3. At least one diagnosis of COPD (ICD9: 491.x, 492.x, 496; ICD10: J41.x, J42, J43.x, J44.x) at any time prior to or on the index date;
- 4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs;
- 5. At least one record in the health insurance system database.

#### • Exclusion criteria:

- 1. Any use of Tio+Olo in free or fixed form within one year prior to the index date. (the free combination will be defined as the prescriptions of the two compounds within 30 days);
- 2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date.

Relevant ICD codes and procedure code are provided in the Annex.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### For other incident LAMA/LABAs combined inhaler cohort

#### Inclusion criteria:

- 1. At least one prescription for LAMA+LABA FDC (Vilanterol/Umeclidinium; Indacaterol /Glycopyrronium) or free combination (LABA: Salmeterol; Formoterol; Procaterol; Indacaterol; Olodaterol, LAMA: Tiotropium bromide; Glycopyrrolate; Umeclidinium) other than Tio/Olo as a new initiation between 1st January 2014 and 31st December 2019 (the free combination will be defined as the prescriptions of the two compounds on the same day);
- 2. Aged ≥ 40 years on the index date (The first dispensing of LAMA+LABA combined inhaler will be defined as the index date);
- 3. At least one diagnosis of COPD at any time prior to or on the index date;
- 4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs;
- 5. At least one record in the health insurance system database.

#### • Exclusion criteria:

- 1. Any use of LAMA+LABA in free or fixed form for one year prior to the index date (the free combination will be defined as the prescriptions of the two compounds within 30 days);
- 2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date.

Relevant ICD codes and procedure code are provided in the Annex.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Figure 1. Patient selection flow chart



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.4 STUDY VISITS

Not applicable.

#### 7. VARIABLES

#### 7.1 EXPOSURES

Exposure of this study is defined as new initiation of Tio/Olo or other LAMA/LABA inhaler (FDC or free combination) during the study period. The free form will be defined as the prescriptions of the two compounds on the same day. Drug codes of interest are provided in the Annex.

#### 7.2 OUTCOMES

#### 7.2.1 Primary outcomes

#### ➤ Incidence rate of adverse events in patients with COPD treated with Tio+Olo

#### List of adverse events:

For acute, potentially recurrent events, including COPD exacerbations listed below, all subjects will be evaluated, regardless of whether such events occurred during the one-year baseline period.

- Respiratory tract disorders
  - 1. Nasopharyngitis
  - 2. Pneumonia
  - 3. COPD exacerbation
- Gastrointestinal disorders
  - 1. Constipation
  - 2. Diarrhoea
- Urinary disorders
  - 1. Urinary retention
  - 2. Urinary tract infection
- Immune system
  - 1. Urticaria

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. Rash

For chronic conditions listed below, subjects who had diagnosis of the condition during the one-year baseline period will be excluded from the incidence of adverse event analysis.

- Cardiovascular disorders
  - 1. Arrhythmia
  - 2. Myocardial ischemia
  - 3. Supraventricular tachycardia
- Ophthalmic disorders
  - 1. Glaucoma
- Serious Adverse Event (SAE)
  - 1. Nonfatal myocardial infarction
  - 2. Nonfatal stroke (hemorrhagic stroke, ischemic stroke and acute cerebrovascular disease)

Lastly, all-cause mortality, a serious adverse event, will be evaluated.

Relevant ICD codes and operational definition are provided in the Annex.

For the analysis of the primary outcome, individuals will be followed up from the index date until the earliest of the following

- 1) Outcome of interest
- 2) disenrollment;
- 3) the end of the study period;
- 4) death;
- 5) discontinuation of the index drug use as a lapse of 45 days without subsequent prescription;
- 6) adding ICS mono on top of Tio/Olo.

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



### 7.2.2 Secondary outcomes

These are not "outcomes" that occurred after the index date in most studies. These are analysis of baseline characteristics of patients who initiated Tio+Olo or other LAMA/LABA.

#### **Basic characteristics:**

• Sex

#### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Age
- Calendar year of cohort entry
- Season of index date (winter, Dec-Feb; spring, Mar-May; summer, Jun-Aug; fall, Sep-Nov)

#### Additional characteristics will be defined during the 1-year pre-index baseline period:

- Specific previous COPD treatments
  - > LAMA monotherapy
  - ➤ LABA monotherapy
  - ➤ ICS monotherapy
  - LAMA/ICS combination therapy on the same day
  - ➤ LAMA+LABA free combinations and fixed dose combination
- Use of other respiratory drugs
  - Mucolytics
  - > Theophylline
  - ➤ Short-acting beta-agonists
  - Short-acting muscarinic antagonists
- Previous acute COPD exacerbation (measured both 12 months and in the 30 days prior to cohort entry), categorized as 0, 1, or 2+.
  - ➤ All exacerbations (Moderate + Severe)
  - An outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections (Moderate); prescriptions within 30 days of each other were considered as continuation of the initial exacerbation.
  - ➤ Hospitalizations or emergency room visits with a primary diagnosis for COPD (Severe); hospitalizations or emergency room visits within 30 days of each other were considered as continuation of the initial exacerbation.
- Hospitalizations caused by exacerbation of COPD in 12 months prior to index date:
  - $\triangleright$  0;
  - **>** 1;
  - >=2:
- All-cause hospitalizations in 12 months prior to index date;
- Comorbidities:
  - > Cardiovascular disease
  - Cerebrovascular disease
  - Diabetes
  - Chronic kidney disease
  - Pneumonia
  - > Cancer
  - Cirrhosis
- Charlson Comorbidity Index (CCI)

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- History of medications dispensed in the 12 months before or on the index date will be identified from the pharmacy dispensing history:
  - > Cardiovascular drugs: antihypertensives, antiarrhythmics, nitrates, heart failure medications
  - > Lipid-lowering medications
  - ➤ Blood glucose-lowering medications
  - Anticoagulants and antiplatelet agents
  - > Antibiotics
  - > Antineoplastic agents

Relevant ICD codes, drugs ATC codes and operational definition are provided in the Annex.



#### 7.3 COVARIATES

Covariates are the same as that listed under 7.2.2.

#### 8. DATA SOURCES

Data sources include Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data. Taiwan Department of Statistics, Ministry of Health and Welfare is the unit designated by the government to manage health and social welfare statistical databases, and to develop data platform for academic research. Through the services provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, researchers may access a wide range of health and welfare data, including claims, mortality (with cause of death) and Taiwan Cancer Registry (TCR). The HWDSC staff encrypt the national ID for all individuals according to a secure encryption algorithm that is not made known to the public. The encrypted ID is unique for all individuals and will be used for linkage between databases.

The ICD-9-CM coding system was used until the end of 2015 and the use of ICD-10-CM codes started on January 1, 2016.

#### 9. DATA MANAGEMENT AND SOFTWARE/TOOLS

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.1 **SOFTWARE/TOOLS**

All analysis will be conducted by SAS software version 9.4 (

#### 9.2 HANDLING OF MISSING VALUES

As administrative data routinely submitted to the health authority, there are no missing value in the health insurance claims. Handling of apparently inconsistent data is described under section 9.3. The small number of subjects with missing information on date of birth or gender will be excluded from the study and described in Figure 1.

#### 9.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

No clinical parameter values (such as blood pressure or laboratory examination results) are available, therefore potential outliers of continuous variables are not a major concern. Apparently inconsistent data, such birth year of 1860 or Tio+Olo prescriptions during the years that it was not covered, would be identified and subjects with inconsistent data will be excluded from analysis and described in Figure 1.

#### 10. DATA ANALYSIS

#### 10.1 MAIN ANALYSIS

All variables, including patient characteristics, baseline measures, and outcomes, will be analyzed descriptively.

- For all analyses, variables will be reported as follows: Continuous variables (e.g., age) will be presented as means (with standard deviation, SD) and/or medians (with interquartile range, IQR), minimum, maximum.
- Categorical variables (e.g., sex) will be presented as absolute and relative frequencies.

We will first describe formation of the study cohort. Patient characteristics at baseline will be described using standard descriptive statistics. Absolute standardized differences (ASDs) will be used to compare the characteristics between the two groups, in which a >0.1 ASD indicates a meaningful difference.

As an objective of the study was to compare the clinical attributes of patients in each study group. The standardized difference will be used as a parameter to quantify the between-group differences for each clinical attribute. This is metric is commonly used in studies utilizing

#### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

secondary health data, in which a standardized difference of larger than 0.1 indicates a meaningful difference with respect to the clinical attribute between the two study groups.

For the analysis of primary outcome, the incidence rates of AEs during entire follow-up period will be calculated based on the following formula:

(Total number of patients in the Tio+Olo cohort experiencing an event of interest for the first time during the given time period) / (Total person-time at risk from current use of Tio+Olo during the given period)

Number of at-risk patients will be defined for specific adverse outcome of interest, taking into account whether it is a chronic condition for which patients with a prevalent condition are not considered at risk.

For the analysis of the primary outcome, individuals will be followed up from the index date until the earliest of the following

- 1) Outcome of interest
- 2) disenrollment;
- 3) the end of the study period;
- 4) death;
- 5) discontinuation of the index drug use as a lapse of 45 days without subsequent prescription;
- 6) adding ICS mono on top of Tio/Olo.

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 10.3 SAFETY ANALYSIS

Not applicable.

#### 11. QUALITY CONTROL

The study will strictly follow relevant BI SOPs. In addition, this study will follow key elements of the Guideline for Good Pharmacoepidemiology Practices (GPP) and the Guideline for Good Pharmacovigilance Practices (GVP).

The statistical analytic approach will be reviewed/repeated by a second analyst to ensure quality control. The study report will be reviewed, approved and archived per BI SOP.

#### 12. REFERENCES

#### 12.1 PUBLISHED REFERENCES

- **R22-0908** Wang C, Xu J, Yang L, et al. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study) a national cross-sectional study. Lancet, 2018, 391(10131): 1706-1717.
- P11-13226 Verhamme KM, Afonso AS, van Noord C, Haag MD, Koudstaal PJ, Brusselle GG, et al. Tiotropium Handihaler and the risk of cardio- or cerebrovascular events and mortality in patients with COPD. Pulm Pharmacol Ther. 2012 Feb;25(1):19-26.
- **R08-1492** Soriano JB, Maier WC, Visick G, Pride NB. Validation of general practitioner-diagnosed COPD in the UK General Practice Research Database. Eur J Epidemiol. 2001;17(12):1075-80.
- **P07-09136** Curkendall SM, Lanes S, de Luise C, et al. Chronic obstructive pulmonary disease severity and cardiovascular outcomes. Eur J Epidemiol. 2006;21(11):803-13.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- **P19-08890** Moretz C, Bengtson LG, Sharpsten L, et al. Evaluation of rescue medication use and medication adherence receiving umeclidinium/vilanterol versus tiotropium bromide/olodaterol. Int J Chron Obstruct Pulmon Dis. 2019 Sep 4;14:2047-2060.
- **P16-05628** Wedzicha J A, et al. Indacaterol–Glycopyrronium versus Salmeterol–Fluticasone for COPD. N Engl J Med, 2016, 2016(374): 2222-2234
- **P07-11820** Wedzicha JA et al. The prevention of COPD exacerbations by salmeterol/fluticasone propionate or tiotropium bromide. Am J Respir Crit Care Med.2008;177:19-26.

#### 12.2 UNPUBLISHED REFERENCES

None

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **ANNEX 1. ADDITIONAL INFORMATION**

# Table 1. Demographic and cohort entry of the Tio/Olo cohort and LAMA/LABA cohort

| | | cohort<br>xxxx | | ABA cohort |
|-------------------------------|---|----------------|---|------------|
| | N | % | N | % |
| Gender | | | | |
| Male | | | | |
| Female | | | | |
| Age | | | | |
| Mean, SD | | | | |
| 40~59 | | | | |
| 60~79 | | | | |
| 80+ | | | | |
| Calendar year of cohort entry | | | | |
| 2014 | | | | |
| 2015 | | | | |
| 2016 | | | | |
| 2017 | | | | |
| 2018 | | | | |
| 2019 | | | | |
| Season of cohort entry date | | | | |
| Spring (Mar-May) | | | | |
| Summer (Jun-Aug) | | | | |
| Fall (Sep-Nov) | | | | |
| Winter (Dec-Feb) | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Table 2. Incidence rate of adverse events in patients with COPD treated with Tio+Olo

| Adverse event | No. of events | Person-Years | Incidence rate<br>(per 100 000<br>person year) | 95% CI |
|---|---|---|---|---|
| Potentially recurrent events | | | | |
| Nasopharyngitis | | | | |
| Pneumonia | | | | |
| Moderate COPD exacerbation | | | | |
| Severe COPD exacerbation | | | | |
| Constipation | | | | |
| Diarrhoea | | | | |
| Urinary retention | | | | |
| Urinary tract infection | | | | |
| Urticaria | | | | |
| Rash | | | | |
| Incident events (no occurrence o | f corresponding | g codes during t | the 1-year baselin | ie period) |
| Arrhythmia | | | | |
| Myocardial ischemia | | | | |
| Supraventricular tachycardia | | | | |
| Glaucoma | | | | |
| Nonfatal myocardial infarction | | | | |
| Nonfatal hemorrhagic stroke | | | | |
| Nonfatal ischemic stroke | | | | |
| Nonfatal Acute, but ill- | | | | |
| defined, cerebrovascular | | | | |
| disease | | | | |
| Death | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Table 3. Secondary outcome (baseline comparison between two study groups)

| - , | | 1 | | | <i>J &amp; 1 )</i> |
|---|---|---|---|---|---|
| | Tio/Ol/ | o cohort | LAM | A/LABA | |
| | | XXXX | со | hort | Standardized |
| | | | N= | XXXX | difference |
| | N | % | N | % | |
| COPD treatments in 1 year prior to inde | ex date | | | | |
| LAMA | | | | | |
| LABA | | | | | |
| ICS | | | | | |
| ICS+LABA free combination | | | | | |
| ICS+LAMA free combination | | | | | |
| LAMA+LABA free combination | | | | | |
| ICS+LAMA+LABA free combination | | | | | |
| ICS/LABA FDC | | | | | |
| LAMA/LABA FDC | | | | | |
| ICS/LAMA/LABA FDC | | | | | |
| Use of other respiratory drugs in 1 year | prior to | index | | | |
| date | | | | | |
| Mucolytics | | | | | |
| Theophylline | | | | | |
| Short-acting beta-agonists (SABA) | | | | | |
| Short-acting muscarinic antagonists | | | | | |
| (SAMA) | | | | | |
| Acute COPD exacerbation in 1 year prior | or to inde | x date | | | |
| Moderate exacerbation | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| Severe exacerbation | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| All exacerbations (Moderate + | | | | | |
| Severe) | | | | | |
| 0 | | | | | |
| 1<br>>=2 | | | | | |
| | c prior to | indov | | | |
| Acute COPD exacerbation in the 30 day date | s prior to | inuex | | | |
| Moderate exacerbation | | | | | |
| 0<br>1 | | | | | |
| >=2 | | | | | |
| Severe exacerbation | | | | | |
| Severe exacerbation | | | | | |

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| | Tio/Olo cohort<br>N=xxxx | | LAM | A/LABA | |
|---|---|---|---|---|---|
| | | | | hort | Standardized |
| | | | N= | XXXX | difference |
| | N | % | N | % | _ |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| All exacerbations (Moderate + | | | | | |
| Severe) | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| Hospitalizations caused by exacerbation | of COPE | in 1 year p | rior to i | ndex date | |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| All-cause hospitalizations in 1 year prior | r to index | date | | | |
| 0 | | | | | |
| 1 | | | | | |
| >=2 | | | | | |
| Comorbidities: | | | | | |
| Cardiovascular disease | | | | | |
| Cerebrovascular disease | | | | | |
| Diabetes | | | | | |
| Chronic kidney disease | | | | | |
| Pneumonia | | | | | |
| Cancer | | | | | |
| Cirrhosis | | | | | |
| Charlson Comorbidity Index (CCI) | | | | | |
| (mean, SD) | | | | | |
| History of medications dispensed in 1 ye | ear prior | to index | | | |
| date | | | | | |
| Cardiovascular drugs: | | | | | |
| Antihypertensives | | | | | |
| Antiarrhythmics | | | | | |
| Nitrates | | | | | |
| Heart failure medications | | | | | |
| Lipid-lowering medications | | | | | |
| Blood glucose–lowering medications | | | | | |
| Anticoagulants and antiplatelet | | | | | |
| agents | | | | | |
| Antibiotics | | | | | |
| Antineoplastic agents | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| Tropricial | ry commucinia. | i iiiioiiiiatioii 🤊 | 9 2022 <b>D</b> 0CIII I | nger mgemem | international O | morr or one or m | ofe of its affiliated c | ompanies |
|---|---|---|---|---|---|---|---|---|

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| Probrietary confidential infort | nation © 2022 Boenringer ing | emeim international Cimbri | or one or more of its affiliated | combanies |
|---|---|---|---|---|

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Appendix 1. Relevant ICD-9/10-CM code and procedure code

| | ICD9 | ICD10 |
|---|---|---|
| For inclusion criteria | | |
| COPD | 491.x, 492.x, 496 | J41.x, J42, J43.x, J44.x |
| For exclusion criteria | | |
| Asthma | 493.x | J45.x |
| Allergic rhinitis | 477.x | J30.x |
| Lung cancer | 162.x | C33.x, C34.x, C7A.090, |
| | | D02.2 |
| Interstitial lung disease | 238.1, 500, 501, 502, 503, | J60, J61, J62.x, J63.x, J64, |
| | 504, 505, 506.4, 508.1, | J65, J66.x, J68.4, J70.x (no |
| | 508.8, 515, 516.x | 70.2), J84.1x (no J84.114), |
| | | J84.2, J84.3, J84.89, J84.9, |
| | | J94.1 |

| <b>Procedure codes</b> | Content |
|---|---|
| 68037A | Lung transplantation |
| 68037B | Lung transplantation - Unilateral lung |
| 68047B | Lung transplantation - bilateral sequential or en bloc double lung |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Appendix 2. List of COPD medication

| Groups | Drug name | ATC code |
|---|---|---|
| LAMA | Tiotropium bromide | R03BB04 |
| | Glycopyrrolate | R03BB06 |
| | Umeclidinium | R03BB07 |
| LABA | Salmeterol | R03AC12 |
| | Formoterol | R03AC13 |
| | Procaterol | R03AC16 |
| | Indacaterol | R03AC18 |
| | Olodaterol | R03AC19 |
| ICS | Beclometasone(=beclomethasone) | R03BA01 |
| | Budesonide | R03BA02 |
| | Fluticasone | R03BA05 |
| | Ciclesonide | R03BA08 |
| ICS/LABA | Salmeterol and Fluticasone | R03AK06 |
| | Formoterol and Budesonide | R03AK07 |
| | Formoterol and Beclometasone | R03AK08 |
| | Vilanterol and Fluticasone furoate | R03AK10 |
| | Formoterol and Fluticasone | R03AK11 |
| LABA/LAMA | Vilanterol and Umeclidinium bromide | R03AL03 |
| | Indacaterol and Glycopyrronium bromide | R03AL04 |
| | Olodaterol and Tiotropium bromide | R03AL06 |
| LABA/LAMA/ICS | Vilanterol, Umeclidinium bromide and Fluticasone furoate | R03AL08 |
| | Formoterol, Glycopyrronium bromide and Beclometasone | R03AL09 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Appendix 3. ICD codes and operational definition of adverse events

| | Adverse events | ICD codes | Operational definition |
|---|---|---|---|
| 1 | Nasopharyngitis | ICD9: 472.2, 460<br>ICD10: J31.1, J00 | Inpatient or outpatient (including ER visit) diagnosis. |
| 2 | Pneumonia | ICD9: 480-486, 487.0<br>ICD10: J10.0, J11.0, J12-<br>J18, | <ol> <li>Primary inpatient diagnosis</li> <li>Inpatient diagnosis.</li> </ol> |
| 3 | Moderate COPD exacerbation | ICD9: 491.x, 492.x, 496<br>ICD10: J41.x, J42, J43.x,<br>J44.x | Outpatient diagnosis plus a prescription for oral corticosteroid or antibiotic for respiratory infection |
| 4 | Severe COPD exacerbation | ICD9: 491.x, 492.x, 496<br>ICD10: J41.x, J42, J43.x,<br>J44.x | Inpatient or ER visits with a primary diagnosis. |
| 5 | Arrhythmia | ICD9: 427.x<br>ICD10: I47.x, I48.x, I49.x | Inpatient or outpatient (including ER visit) diagnosis. |
| 6 | Myocardial ischemia | ICD9: 410.x, 411.x, 413.x<br>ICD10: I20.x, I21.x, I22.x,<br>I23.x, I24.x | Inpatient or outpatient (including ER visit) diagnosis. |
| 7 | Supraventricular tachycardia | ICD9: 427.0<br>ICD10: I47.1 | Inpatient or outpatient (including ER visit) diagnosis. |
| 8 | Constipation | ICD9: 564.0, 564.00,<br>564.09<br>ICD10: K59.0, K59.00,<br>K59.09 | Inpatient or outpatient (including ER visit) diagnosis. |
| 9 | Diarrhoea | ICD9: 787.91<br>ICD10: R19.7 | Inpatient or outpatient (including ER visit) diagnosis. |
| 10 | Urinary retention | ICD9: 788.2, 788.20,<br>788.29<br>ICD10: R33.x | Inpatient or outpatient (including ER visit) diagnosis. |
| 11 | Urinary tract infection | ICD9: 590, 595, 601, 604<br>ICD10: N10, N12, N15.1,<br>N30.0, N30.8, N30.9,<br>N41.0, N41.2, N41.3,<br>N39.0 | <ol> <li>Primary inpatient diagnosis</li> <li>Inpatient diagnosis.</li> <li>Either inpatient diagnosis or at least 2 outpatients (including ER visit) diagnosis; diagnostic interval within 30 days.</li> </ol> |
| 12 | Urticaria | ICD9: 708.x<br>ICD10: L50.x | Inpatient or outpatient (including ER visit) diagnosis. |
| 13 | Rash | ICD9: 782.1<br>ICD10: R21 | Inpatient or outpatient (including ER visit) diagnosis. |

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| 14 | Glaucoma | ICD9: 365.x | Inpatient or outpatient |
|---|---|---|---|
| | | ICD10: H40.x | (including ER visit) diagnosis |
| | | | from ophthalmologist. |
| 15 | Nonfatal myocardial | ICD9: 410.x, 411.x | 1. Primary inpatient diagnosis |
| | infarction | ICD10: I21.x, I22.x, I23.x | + hospital discharge |
| | | | without death certificates |
| | | | 2. Inpatient diagnosis + |
| | | | hospital discharge without |
| | | | death certificates |
| 16 | Nonfatal hemorrhagic stroke | ICD9: 430, 431, 432.x | 1. Primary inpatient diagnosis |
| | | ICD10: 160.x, 161.x, 162.x | + hospital discharge |
| | | | without death certificates |
| | | | 2. Inpatient diagnosis + |
| | | | hospital discharge without |
| | | | death certificates |
| 17 | Nonfatal ischemic stroke | ICD9: 433.x, 434.x | 1. Primary inpatient diagnosis |
| | | ICD10: 163.x, 166.x | + hospital discharge |
| | | | without death certificates |
| | | | 2. Inpatient diagnosis + |
| | | | hospital discharge without |
| | | | death certificates |
| 18 | Nonfatal acute | ICD9: 436 | 1. Primary inpatient diagnosis |
| | cerebrovascular disease | ICD10: 167.8 | + hospital discharge |
| | | | without death certificates |
| | | | 2. Inpatient diagnosis + |
| | | | hospital discharge without |
| | | | death certificates |
| 19 | Fatal events | | All cause of death |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Appendix 4. ICD codes and operational definition of comorbidities

| | Comorbidities: | ICD codes | Operational definition |
|---|---|---|---|
| 1. | Diabetes | ICD9: 250 | Either inpatient diagnosis or |
| | | ICD10: E10.x-E11.x | more than twice outpatient |
| | | | diagnosis |
| 2. | Cardiovascular disease | ICD9: 250.7, 401-405, | Either inpatient diagnosis or |
| | | 410-414, 425-428, 429.1- | more than twice outpatient |
| | | 429.3, 441, 442, 458 | diagnosis |
| | | ICD10: E10.5x, E11.5x, | |
| | | 110-113.x, 115.x, 120.x- | |
| | | 122.x, 124.x, 125.x, 142.x- | |
| | | 144, 145.xx, 146.x-149.x, | |
| | | I50.xx, I51.5, I51.7, I51.9, | |
| | | 171.xx, 179.0, 172.x, | |
| | | 177.7x, 195.x | |
| 3. | Cerebrovascular disease | ICD9: 430-438 | Either inpatient diagnosis or |
| | | | more than twice outpatient |
| | | 166.x, G45.x, G46.x, 167.x- | diagnosis |
| | | 169.x | |
| 4. | Cancer | ICD9: 140-199, 200-208 | Inpatient diagnosis. |
| | | ICD10: C00-C26, C30-34, | |
| | | C37-39, C40-41, C43-49, | |
| | | C4A, C50-58, C60-69, | |
| | | С70-79,С7А, С7В, С80- | |
| | | 86, C88, C90-96, | |
| 5. | Chronic kidney disease | ICD9: 585-587, | Either inpatient diagnosis or |
| | | ICD10: N18-19, N26.1, | more than twice outpatient |
| | | N26.9 | diagnosis |
| 6. | Pneumonia | ICD9: 480-486, 487.0 | Inpatient diagnosis |
| | | ICD10: J10.0, J11.0, J12- | |
| | | J18, | |
| 7. | Cirrhosis | | Either inpatient diagnosis or |
| | | ICD10: K70.3x, K74.3, | more than twice outpatient |
| | | K74.4, K74.5, K74.6x | diagnosis |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Appendix 5. Drugs of interest

| Groups | ATC code |
|---|---|
| Use of other respiratory drugs | |
| Mucolytics | R05CB, R05CB01, R05CB02, R05CB03, R05CB04, R05CB05, |
| | R05CB06, R05CB10, R05CB11, R05CB91, R05CB92 |
| Theophylline | R03DA04, R03DA54, R03DA74, R03DB04 |
| SABA | R03AC02, R03AC03, R03AC04, R03AC06 |
| SAMA | R03BB01 |
| SABA/SAMA | R03AL01, R03AL02 |
| Drugs for COPD exac | cerbation treatment |
| Oral corticosteroid | H02AB01, H02AB02, H02AB04, H02AB05, H02AB06, H02AB08, |
| | H02AB10, H02BX, H02BX91 |
| Antibiotic for COPD | J01AA02, J01CA04, J01CR02, J01CR05, J01EE01, J01DC01, |
| exacerbation | J01DC02, J01DC03, J01DC04, J01DC05, J01DC06, J01DC07, |
| | J01DC09, J01DC14, J01DD01, J01DD02, J01DD04, J01DD05, |
| | J01DD06, J01DD07, J01DD08, J01DD12, J01DD13, J01DD14, |
| | J01DD52, J01DD62, J01DE01, J01DE02, J01FA01, J01EA02, |
| | J01EA03, J01EA06, J01EA07, J01EA08, J01FA09, J01FA10, |
| | J01FA15, J01FA91, J01MA01, J01MA02, J01MA03, J01MA04, |
| | J01MA06, J01MA07, J01MA09, J01MA12, J01MA14, J01MA15 |
| Drugs for Medication | history |
| • Cardiovascular o | lrugs |
| Anti-hypertensives | C02AA01, C02AA02, C02AA04, C02AB01, C02AB02, C02AC01, |
| | C02CA01, C02CA04, C02CA, C02CC02, C02DA01, C02DB02, |
| | C02DC01, C02DD01, C02LA01, C02LA50, C02LA51, C02LB01, |
| | C02LG02, C02N, C03AA01, C03AA03, C03AA06, C03AA07, |
| | C03AA, C03BA04, C03BA08, C03BA11, C03CA01, C03CA02, |
| | C03CA04, C03CC01, C03DA01, C03DA04, C03DB01, C03DB02, |
| | C03EA01, C03EA, C07AA01, C07AA02, C07AA03, C07AA05, |
| | C07AA06, C07AA07, C07AA12, C07AA15, C07AA19, C07AB02, |
| | C07AB03, C07AB04, C07AB05, C07AB07, C07AB09, C07AB12, |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| 1 7 | 0074 C01 |
|---|---|
| | C07AG01, C07AG02, C07BA68, C07BB02, C07CA03, C07CB03, |
| | C07DA06, C08CA01, C08CA02, C08CA03, C08CA04, C08CA05, |
| | C08CA07, C08CA08, C08CA09, C08CA12, C08CA13, C08CA15, |
| C08DA01, C08DB01, C09AA01, C09AA02, C09AA03, C | |
| | C09AA05, C09AA06, C09AA07, C09AA08, C09AA09, C09AA16, |
| | C09BA01, C09BA02, C09BA04, C09BB04, C09BB05, C09BB, |
| | C09BB, C09CA01, C09CA02, C09CA03, C09CA04, C09CA06, |
| | C09CA07, C09CA08, C09CA09, C09DA01, C09DA03, C09DA04, |
| | C09DA06, C09DA07, C09DA08, C09DA09, C09DB01, C09DB02, |
| | C09DB04, C09DB07, C09DX01, C09DX03, C09DX04, C09XA02, |
| | C09XA52, C09XA53, C09XA54 |
| Antiarrhythmics | C01AA04, C01AA05, C01AA07, C01AA08, C01AB01, C01AC01, |
| | C01BA01, C01BA02, C01BA03, C01BA04, C01BA08, C01BB01, |
| | C01BB02, C01BC03, C01BC04, C01BD01, C01BD07, C01CA02, |
| | C01CA04, C01CA06, C01EB10, C01EB17, C07AA01, C07AA02, |
| | C07AA03, C07AA05, C07AA07, C07AA12, C07AA15, C07AA |
| | C07AB02, C07AB03, C07AB04, C07AB05, C07AB07, C07AB09, |
| | C07AB12, C08DA01, C08DB01 |
| Heart failure | C01AA04, C01AA05, C01AA07, C01AA08, C01AB01, C01AC01, |
| medications | C01CA02, C01CA07, C01CE02, C01EB09, C01EB17, C03CA02, |
| | C03CA04, C03DA04, C07AG02, C09AA01, C09AA02, C09AA03, |
| | C09AA04, C09AA05, C09AA06, C09AA07, C09AA08, C09AA09, |
| | C09AA16, C09CA01, C09CA02, C09CA03, C09CA04, C09CA06, |
| | C09CA07, C09CA08, C09CA09 |
| Nitrates | C01DA02, C01DA05, C01DA08, C01DA14 |
| Lipid-lowering | medications |
| Lipid Modifying | C10AA01, C10AA02, C10AA03, C10AA04, C10AA05, C10AA07, |
| Agents, Plain C10AA08, C10AB01, C10AB02, C10AB03, C10AB04, C | |
| C10AB06, C10AB09, C10AC01, C10AC02, C10AC03, C10A | |
| | C10AD02, C10AD03, C10AD06, C10AD, C10AX02, C10AX09, |
| | C10AX13, C10AX14, C10AX |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| Lipid Modifying | C10BA01, C10BA02, C10BA03, C10BA05, C10BX03 |
|---|---|
| Agents, Combinations | |
| Blood glucose-lowering medications | |
| Insulins and analogues | A10AB01, A10AB03, A10AB04, A10AB05, A10AB06, A10AB30, |
| | A10AC01, A10AC03, A10AC30, A10AD01, A10AD03, |
| | A10AD04, A10AD05, A10AD06, A10AE01, A10AE04, A10AE05, |
| | A10AE06, A10AE54 |
| | A10BA02, A10BA03, A10BB01, A10BB02, A10BB03, A10BB04, |
| drugs, excl. insulins | A10BB05, A10BB07, A10BB08, A10BB09, A10BB12, A10BB31, |
| | A10BD02, A10BD03, A10BD05, A10BD07, A10BD08, A10BD09, |
| | A10BD10, A10BD11, A10BD13, A10BD14, A10BD, A10BD15, |
| | A10BD19, A10BD20, A10BD21, A10BD24, A10BF01, A10BF02, |
| | A10BG02, A10BG03, A10BH01, A10BH02, A10BH03, A10BH04, |
| | A10BH05, A10BJ01, A10BJ02, A10BJ03, A10BJ05, A10BJ06, |
| | A10BK01, A10BK02, A10BK03, A10BK04, A10BX01, A10BX02, |
| | A10BX03, A10BX08 |
| Anticoagulants an | d antiplatelet agents |
| Vitamin K antagonists | B01AA02, B01AA03 |
| Heparin group | B01AB01, B01AB04, B01AB05, B01AB06, B01AB10 |
| Platelet aggregation | B01AC04, B01AC05, B01AC06, B01AC07, B01AC09, B01AC11, |
| inhibitors excl. heparin | B01AC13, B01AC16, B01AC17, B01AC21, B01AC22, B01AC23, |
| | B01AC24, B01AC27, B01AC30 |
| Enzymes | B01AD01, B01AD02, B01AD04, B01AD10, B01AD11 |
| Direct thrombin | B01AE07 |
| inhibitors | |
| Direct factor Xa | B01AF01, B01AF02, B01AF03 |
| inhibitors | |
| Other antithrombotic | B01AX05 |
| agents | |
| • Antibiotic | 1 |
| L | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| Antibacterials for | J01AA01, J01AA02, J01AA03, J01AA04, J01AA06, J01AA07, |
|---|---|
| systemic use | J01AA08, J01AA09, J01AA12, J01AA56, J01BA01, J01BA02, |
| | J01BA51, J01CA01, J01CA02, J01CA03, J01CA04, J01CA06, |
| | J01CA08, J01CA09, J01CA10, J01CA12, J01CA13, J01CA14, |
| | J01CA15, J01CA16, J01CA18, J01CA20, J01CA91, J01CE01, |
| | J01CE02, J01CE08, J01CE09, J01CE30, J01CF01, J01CF02, |
| | J01CF04, J01CF05, J01CG01, J01CR01, J01CR02, J01CR03, |
| | J01CR04, J01CR05, J01CR50, J01CR50, J01CR50, J01DB01, |
| | J01DB02, J01DB03, J01DB04, J01DB05, J01DB06, J01DB07, |
| | J01DB08, J01DB09, J01DC01, J01DC02, J01DC03, J01DC04, |
| | J01DC05, J01DC06, J01DC07, J01DC09, J01DC14, J01DD01, |
| | J01DD02, J01DD04, J01DD05, J01DD06, J01DD07, J01DD08, |
| | J01DD12, J01DD13, J01DD14, J01DD52, J01DD62, J01DE01, |
| | J01DE02, J01DF01, J01DH02, J01DH03, J01DH04, J01DH51, |
| | J01DI02, J01DI54, J01E, J01EA01, J01EB01, J01EB02, J01EB05, |
| | J01EB06, J01EB20, J01EC, J01EC01, J01EC02, J01EC20, |
| | J01ED01, J01ED05, J01ED20, J01EE01, J01FA01, J01EA02, |
| | J01EA03, J01EA06, J01EA07, J01EA08, J01FA09, J01FA10, |
| | J01FA15, J01FA91, J01FF01, J01FF02, J01GA01, J01GB01, |
| | J01GB03, J01GB04, J01GB05, J01GB06, J01GB07, J01GB08, |
| | J01GB09, J01GB11, J01MA01, J01MA02, J01MA03, J01MA04, |
| | J01MA06, J01MA07, J01MA09, J01MA12, J01MA14, J01MA15, |
| | J01MB01, J01MB02, J01MB03, J01MB04, J01MB08, J01RA02, |
| | J01XA01, J01XA02, J01XB, J01XB01, J01XC01, J01XD01, |
| | J01XD02, J01XD03, J01XE, J01XE01, J01XE02, J01XX01, |
| | J01XX04, J01XX05, J01XX07, J01XX08, J01XX09, J01XX91 |
| Antimycotics for | J02AA01, J02AB01, J02AB02, J02AC01, J02AC02, J02AC03, |
| systemic use | J02AC04, J02AC05, J02AX01, J02AX04, J02AX05, J02AX06 |
| Antimycobacterials | J04AA03, J04AB01, J04AB02, J04AB03, J04AB04, J04AB91, |
| | J04AC01, J04AC51, J04AD01, J04AK01, J04AK02, J04AK04, |
| | J04AM02, J04AM03, J04AM05, J04AM06, J04AM07, J04BA01, |
| | J04BA02 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template

c40431892-01 

| Antineoplastic age | ents |
|---|---|
| Alkylating agents | L01AA01, L01AA02, L01AA03, L01AA06, L01AA09, L01AB01, |
| | L01AC01, L01AC03, L01AD01, L01AD02, L01AD06, L01AX03, |
| | L01AX04 |
| Antimetabolites | L01BA01, L01BA04, L01BA05, L01BB02, L01BB03, L01BB04, |
| | L01BB05, L01BB06, L01BC01, L01BC02, L01BC03, L01BC05, |
| | L01BC06, L01BC07, L01BC53, L01BC59 |
| Plant alkaloids and | L01CA01,L01CA02, L01CA04, L01CB01, L01CD01, L01CD02, |
| other natural products | L01CE01, L01CE02 |
| Cytotoxic antibiotics | L01DA01, L01DB01, L01DB02, L01DB03, L01DB04, L01DB06, |
| and related substances | L01DB07, L01DC01, L01DC03, L01DC04 |
| Protein kinase inhibitors | L01EA01, L01EA02, L01EA03, L01EA05, L01EB01, L01EB02, |
| | L01EB03, L01EB04, L01EB07, L01EC01, L01EC02, L01ED01, |
| | L01ED02, L01ED03, L01ED04, L01ED05, L01EE01, L01EF01, |
| | L01EF02, L01EG01, L01EG02, L01EH01, L01EJ01, L01EK01, |
| | L01EL01, L01EM02, L01EX01, L01EX02, L01EX03, L01EX04, |
| | L01EX05, L01EX07, L01EX08, L01EX09, L01EX10, L01EX14 |
| Other antineoplastic | L01XA01, L01XA02, L01XA03, L01XB01, L01XC02, L01XC03, |
| agents | L01XC06, L01XC07, L01XC08, L01XC12, L01XC13, L01XC14, |
| | L01XC15, L01XC17, L01XC18, L01XC19, L01XC21, L01XC24, |
| | L01XC26, L01XC31, L01XC32, L01XF01, L01XG01, L01XG02, |
| | L01XG03, L01XK01, L01XK04, L01XX02, L01XX05, L01XX11, |
| | L01XX23, L01XX27, L01XX35, L01XX41, L01XX52, L01XX |
| Hormones and related | L02AA01, L02AA91, L02AB01, L02AB02, L02AE01, L02AE02, |
| agents | L02AE03, L02AE04 |
| Hormone antagonists | L02BA01, L02BA02, L02BB01, L02BB03, L02BB04, L02BB05, |
| and related agents | L02BG01, L02BG03, L02BG04, L02BG06, L02BX02, L02BX03 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) Template c40431892-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals **prior to approval**.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| TSTAT<br>(for NISnd only) | X | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

**Study Title:** Safety profile of Tiotropium + Olodaterol used as maintenance treatment in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data

**Study Number:** 1237-0109

Name/Date:

**Protocol Version:** 1.0

Position:

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| | | • |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |

Signature: